CLINICAL TRIAL: NCT07395609
Title: High Frequency Stimulation to Improve Cognition, Mobility, and Affect in Individuals With Subjective Cognitive Decline
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB202500587
Record Dates: First submitted 2025-09-10; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Subjective Cognitive Decline (SCD); Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): Participants in this group will receive white noise sensory stimulation rather than a constant flicker frequency.
  Interventions: Behavioral: Sham White Noise Stimulation
- Flicker Stimulation (Experimental): Participants in this group will receive sensory visual plus auditory flicker stimulation.
  Interventions: Behavioral: Flicker Stimulation

INTERVENTIONS:
Behavioral: Flicker Stimulation — Investigators will combine ultrasound (≥22 kHz) and near-infrared two-photon stimulation (890-940 nm) to deliver rhythmic input in a subliminal, comfortable manner, without the side effects associated with visible flicker.
  Arms: Flicker Stimulation
Behavioral: Sham White Noise Stimulation — The control group will receive white noise sensory stimulation rather than a constant flicker frequency.
  Arms: Control

SUMMARY:
The goal is to determine whether three months of at least three times / week of sensory flicker stimulation improves cognition, mobility, and affect in older adults with Subjective Cognitive Decline (SCD), relative to an SCD control group receiving white noise sensory stimulation. Investigators will also determine whether the intervention slows cortical thinning and declines in brain functional network segregation and changes in blood biomarkers of Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and women 65-89 years old
* Ability to walk unassisted for 10 min
* English speaking

Additional Inclusion Criteria for SCD:

* No evidence of dementia or MCI based on cognitive screening (i.e., Montreal Cognitive Assessment (MoCA) score within normal limits for age, education, and sex using the NACC Uniform Data Set (UDS) norms8
* Global Clinic Dementia Rating (CDR) score must be 0 or 0.531
* Subjective report of cognitive complaints with scores >20 on the Cognitive Change Index (CCI-20), a validated scale of subjective cognitive decline6; this scale consists of 20 items that are rated on a 5-point Likert scale, where 1= "Normal: No change compared to 5 years ago", 3= "Mild Problem: Some change compared to 5 years ago) and 5="Severe Problem: Much worse compared to 5 years ago"
* Family history of dementia/probable AD in first degree relative (parents, children, siblings)
* Normal functional behavior in terms of daily activities, based on the Functional Activities Scale32
* In line with recommendations of the SCD task force33 an informant must be available for two reasons: a) to provide information about the participant's cognition using the informant version of the CDR and CCI-20, and b) to corroborate normal IADL's on the Functional Activity Questionnaire32 (informant data will be collected via a phone call and linked by code with the participant data).

Exclusion Criteria:

* If participants score less than 21 on the Telephone Interview for Cognitive Status (TICS)
* Significant medical event requiring hospitalization in the past 6 months that has the potential to contaminate data being collected (fracture, hospitalization etc.)
* Severe visual impairment or corrected visual acuity less than 20/40, which would preclude completion of assessments
* Inability to undergo MRI brain imaging due to claustrophobia or implants such as pacemakers, heart valves, brain aneurysm clips, orthodontics, certain non-removable body jewelry, or shrapnel containing ferromagnetic metal
* History of severe stroke
* Any major ADL disability (unable to feed, dress, bath, use the toilet, or transfer)
* Report of lower extremity pain due to osteoarthritis that significantly limits mobility
* Diagnosis or treatment for rheumatoid arthritis
* Known neuromuscular disorder or overt neurological disease (e.g. Multiple Sclerosis, Rhabdomyolysis, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, Parkinson's Disease, ALS etc.)
* Unable to communicate because of severe hearing loss or speech disorder
* Planned surgical procedure or hospitalization in the next 4 months (joint replacement, coronary artery bypass graft, etc.)
* Severe pulmonary disease, requiring the use of supplemental oxygen
* Terminal illness, as determined by a physician
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Use of walker or wheelchair

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  Investigators will comprehensively assess behavior at three times (baseline, half-way through (1.5 months), and after the intervention (3months)) using the NIH Toolbox. Composite Scores of Fluid Cognition from the Cognition Toolbox will serve as primary metrics for cognition.
Grip strength | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  Participants will grip a machine which measures their grip strength in kg.
10m Gait Speed | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  Participants will walk unassisted for 10 meters. Their speed will be measured in seconds.
Clinical Test of Sensory Interaction on Balance (CTSIB) | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  Participants will, with eyes open and closed, walk on rough and smooth terrain. Investigators will measure sway area (measured in m^2/s^4).
Affect - POMS-2 | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  This test is used to assess transient feelings and mood among individuals aged 13 years and above.
  Scoring:
  0 - Not at all
  1. - A little
  2. - Moderately
  3. - Quite a Lot
  4. - Extremely
  Except "Relaxed" and "Efficient", and they score the reverse:
Affect - Ryff Scales of Psychological Wellbeing | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  Respondents agree or disagree with 42 statements using a 6-point scale (1 = strongly agree; 6 = strongly disagree).
Affect - Satisfaction with Life Scale | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  The possible range of scores is 5-35. Scores between 5-9 indicate the respondent is extremely dissatisfied with life, whereas scores between 31-35 indicate the respondent is extremely satisfied.
Affect - Perceived Stress Scale | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  Score is obtained by reverse-scoring items 4, 5, 7, and 8 and then summing the scores.
Affect - Apathy Evaluation Scale | Baseline, halfway through (1.5 months), and post-intervention (3 months)
  After recoding all necessary items, sum up all scores.
Brain Structure and Network Function | Baseline, and post-intervention (3 months)
  Investigators will assess brain structure via a T1 MRI to measure cortical thickness in dorsolateral prefrontal, sensorimotor, and insular cortices using the CAT computational anatomy toolbox; brain network function via resting-state fMRI to capture functional segregation of dorsolateral prefrontal, sensorimotor, and insular networks (subserving cognition, mobility, and affect respectively) using the CONN toolbox.
Blood-based AD pathology (Aβ17) | Baseline, and post-intervention (3 months)
  Investigators will assess levels of Aβ17 [units], which is sensitive to AD. Blood samples will be processed on campus by UF's Florida Alzheimer's Disease Research Center Biomarker Core. Blood will be centrifuged and placed into -80°C storage maintained by the PIs. Coded blood samples will be analyzed in the final year of this project. These biomarker levels will not be shared with participants, as this is not a diagnostic laboratory.
Blood-based AD pathology [p-tau] | Baseline, and post-intervention (3 months)
  Investigators will assess levels of p-tau [units], which is sensitive to AD. Blood samples will be processed on campus by UF's Florida Alzheimer's Disease Research Center Biomarker Core. Blood will be centrifuged and placed into -80°C storage maintained by the PIs. Coded blood samples will be analyzed in the final year of this project. These biomarker levels will not be shared with participants, as this is not a diagnostic laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Seidler, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States